CLINICAL TRIAL: NCT04307316
Title: Effects of Active Cycle of Breathing Technique on Pulmonary Functions After CABG During Phase 1 Cardiac Rehabilitation
Brief Title: Effects of ACBT on Pulmonary Function After CABG During Phase 1 Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00423 Nouman Hussain
Record Dates: First submitted 2020-03-06; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: Active cycle of breathing technique; Chest expansion; Coronary artery bypass graft surgery; FEV1; FVC; PEFR

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACBT group (Experimental): Active cycle breathing technique
  Interventions: Other: ACBT group
- Conventional treatment group (Active Comparator): Conventional treatment group
  Interventions: Other: Conventional Physical therapy

INTERVENTIONS:
Other: ACBT group — ACBT:
  Breathing control 3 to 4 Thoracic Expansion Exercise A: 3 seconds hold B: Chest clapping C: Chest vibration Forced Expiratory Technique Breathing control A: 3 seconds hold B: Chest clapping C: Chest vibration 3 to 4 Thoracic Expansion Exercise Breathing control 1-2 Huff combine with breathing control Huff and cough
  Chest Physical Therapy Early mobilization
  Arms: ACBT group
Other: Conventional Physical therapy — Chest percussion, deep breathing, Huff and cough. Early mobilization
  Arms: Conventional treatment group

SUMMARY:
This study is designed to determine the effects of Active cycle of breathing technique (ACBT) on cardiopulmonary parameters of post CABG patients. A randomized control trial was conducted with a sample size of 40 post CABG patients. Non probability Convenience Sampling Technique was used to collect sample and randomization was done through sealed envelope method to allocate participants to the groups. Patients in experimental group did ACBT along with the conventional treatment protocol that was performed in the control group. Subjects completed the exercise protocol of 5 days. Both male and female post CABG patients of age 30-65 years who were vitally stable were included in study. Data was analyzed on Statistical Package for the Social Sciences (SPSS) version 21. Normality was assessed through shapiro wilk test. Parametric tests were applied on normally distributed variables and non parametric tests were applied for the non normally distributed data. Confidence interval was kept at 95% and p value <0.05 was considered significant.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) is a surgery in which new routes are created around narrow and blocked coronary arteries, that allow proper flow of blood to provide oxygen and nutrients to the heart muscles. The grafts used in CABG can be a vein from lower extremity or any artery of chest. CABG is a surgery in which obstructed coronary arteries are replaced with autologous arteries and veins used as implant, which are fully or moderately congested by atherosclerotic plaque. ACBT is a method used to clear out the secretion from the chest. The purpose of ACBT treatment is to remove secretions from the chest that helps to reduce the frequency of infection, which control the additional airway impairment and worsening the lungs functions that may help in reducing the rate of progress of lung disease. After CABG surgery respiratory therapy is used rationally to inhibit the post-operative complications. Respiratory physiotherapy is routinely used in the prevention and treatment of post-operative pulmonary complications after cardiac surgery. The ultimate goal of physiotherapy in CABG patient is to improve increase lung volume, prevent atelectasis, enhance ventilation-perfusion matching, to increase sputum clearance, and decrease pain. ACBT technique can perform independently by patient with about applying manual technique. ACBT is very effective to improve oxygen saturation, control respiratory rate, and chest clearance after major surgeries. The efficiency of ACBT treatment has been checked out in stable cystic fibrosis, Chronic obstructive pulmonary disease and abdominal surgery. However, there is limited literature related to its use in patients after CABG surgery. The purpose of this research was to examine the effect of ACBT versus conventional chest physiotherapy after CABG surgery.

In 2018 a study was conducted on effect of ACBTs in post coronary artery bypass grafting patient and he concluded that ACBTs technique is a better way of treatment in coronary artery bypass grafting surgery patients. The determination of this research was to calculate the effectiveness of ACBT in CABG surgery patients. In this study total 15 patients were involved. All the patients were checked out by visual analogue scale for pain, 6-minute walk test (6MWT) for endurance and chest expansion was also measured. It concluded that chest expansion and 6MWT was improved in both groups.

ACBT is an effective technique implemented by the patient to secrete out the sputum from the main airway. The ACBT technique is combined breathing maneuvers to advance the efficiency of cough, untie and clear the secretions and increase the ventilation.

In 2016 a study was conducted observed the effects of ACBTs in post CABG surgery patients and The ACBTs treatment decrease the intensity of pulmonary impairments in post abdominal surgery.There is limited data available in support of effects of ACBTs on pulmonary functions after CABG surgery.

In 2015 a study was conducted to evaluate the effects of ACBTs on chest expansion, arterial blood gases, oxygen saturation, blood pressure, respiratory rate and other vitals in Chronic Obstructive Pulmonary disease (COPD) patients during 1st phase of cardiac rehab after CABG surgery. It concluded that ACBT are much effective than routine physiotherapy protocol in patients who have gone under coronary artery bypass grafting.

The present study is intended to observe the effects of ACBT on pulmonary function including lung volumes and capacities, chest expansion as well as the vitals of post operative CABG patients undergoing phase 1 cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Vitally stable post CABG patients

Exclusion Criteria:

* Hemodynamically unstable patients
* Patient after re-opening of sternum.
* Infected patients
* Patients who cannot speak Urdu, Punjabi or English language.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | After 5days
  Forced Expiratory Volume in 1 second (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
Forced vital capacity (FVC) | After 5days
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
FEV1/FVC | After 5days
  FEV1/FVC measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65).
Peak expiratory flow rate (PEFR) | After 5days
  Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
Chest expansion | After 5 days
  Chest expansion at xiphoid level measured by finding the difference in measurements during inhalation and exhalation.

SECONDARY OUTCOMES:
Heart rate | After 5days
  Heart rate is measured as part of vitals through heart rate monitor.
Respiratory rate | After 5 days
  Respiratory rate as part of vitals standing at bedside of the patients
Systolic and diastolic blood pressure | After 5days
  Blood pressure is measured through sphygmomanometer
Oxygen Saturation (SPO2) | After 5days
  Oxygen saturation measured through pulse oximeter as part of vitals

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bachar BJ, Manna B. Coronary Artery Bypass Graft. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507836/ PMID 29939613
- [Background] Freitas ER, Soares BG, Cardoso JR, Atallah AN. Incentive spirometry for preventing pulmonary complications after coronary artery bypass graft. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD004466. doi: 10.1002/14651858.CD004466.pub3. PMID 22972072
- [Background] Hue B, Pelhate M, Callec JJ, Chanelet J. Synaptic transmission in the sixth ganglion of the cockroach: action of 4-aminopyridine. J Exp Biol. 1976 Dec;65(3):517-27. doi: 10.1242/jeb.65.3.517. PMID 190333
- [Background] Zanini M, Nery RM, de Lima JB, Buhler RP, da Silveira AD, Stein R. Effects of Different Rehabilitation Protocols in Inpatient Cardiac Rehabilitation After Coronary Artery Bypass Graft Surgery: A RANDOMIZED CLINICAL TRIAL. J Cardiopulm Rehabil Prev. 2019 Nov;39(6):E19-E25. doi: 10.1097/HCR.0000000000000431. PMID 31343586
- [Background] Uzmezoglu B, Altiay G, Ozdemir L, Tuna H, Sut N. The Efficacy of Flutter(R) and Active Cycle of Breathing Techniques in Patients with Bronchiectasis: A Prospective, Randomized, Comparative Study. Turk Thorac J. 2018 Jul;19(3):103-109. doi: 10.5152/TurkThoracJ.2018.17050. Epub 2018 Jun 12. PMID 30083399
- [Background] Lewis LK, Williams MT, Olds TS. The active cycle of breathing technique: a systematic review and meta-analysis. Respir Med. 2012 Feb;106(2):155-72. doi: 10.1016/j.rmed.2011.10.014. Epub 2011 Nov 18. PMID 22100537
- [Background] Thybo Karanfil EO, Moller AM. Preoperative inspiratory muscle training prevents pulmonary complications after cardiac surgery - a systematic review. Dan Med J. 2018 Mar;65(3):A5450. PMID 29510803
- [Background] Renault JA, Costa-Val R, Rosseti MB, Houri Neto M. Comparison between deep breathing exercises and incentive spirometry after CABG surgery. Rev Bras Cir Cardiovasc. 2009 Apr-Jun;24(2):165-72. doi: 10.1590/s0102-76382009000200012. PMID 19768295
- [Background] Filbay SR, Hayes K, Holland AE. Physiotherapy for patients following coronary artery bypass graft (CABG) surgery: limited uptake of evidence into practice. Physiother Theory Pract. 2012 Apr;28(3):178-87. doi: 10.3109/09593985.2011.582231. Epub 2011 Aug 8. PMID 21823991